CLINICAL TRIAL: NCT03206073
Title: A Phase I/II Study of Pexa-Vec Oncolytic Virus in Combination With Immune Checkpoint Inhibition in Refractory Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170092; 17-C-0092
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Adenocarcinoma; Refractory Cancer; Colorectal Neoplasms
Keywords: Oncolytic Vaccinia Virus; Tumor Cell Death; Viral Therapy; Anti-Tumor Immunity
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1/Arm A1 Pexa-Vec + Durvalumab (Experimental): Pexa-Vec escalation dose levels + Durvalumab
  Interventions: Drug: Durvalumab; Biological: Pexa-Vec
- 2/Arm A2 Pexa-Vec +Durvalumab (Experimental): Maximum tolerated dose (MTD) of Pexa-Vec after the MTD is established +Durvalumab
  Interventions: Drug: Durvalumab; Biological: Pexa-Vec
- 3/Arm B1 Pexa-Vec + Durvalumab +Tremelimumab (Experimental): Pexa-Vec escalation dose levels + Durvalumab +Tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Biological: Pexa-Vec
- 4/Arm B2 (Experimental): MTD of Pexa-Vec after the MTD is established+Durvalumab + Tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Biological: Pexa-Vec

INTERVENTIONS:
Drug: Durvalumab — 1500 mg of durvalumab via intravenous (IV) infusion on Day 1 of each cycle until patients meet off treatment criteria
  Other Names: MEDI-4736
Drug: Tremelimumab — 300 mg of tremelimumab via intravenous (IV) infusion on Day 1 of cycle 1
  Other Names: CP-675,206
  Arms: 3/Arm B1 Pexa-Vec + Durvalumab +Tremelimumab; 4/Arm B2
Biological: Pexa-Vec — 3 x 10E^8 plaque-forming unit (pfu) (Dose Level (DL) 1) via intravenous (IV) infusion for 4 doses: Day 12, Day 2, Day 16 of Cycle 1 and Day 2 of Cycle 2.
  Other Names: Pexa-Vec, INN pexastimogene devacirepvec
  Arms: 1/Arm A1 Pexa-Vec + Durvalumab; 3/Arm B1 Pexa-Vec + Durvalumab +Tremelimumab
Biological: Pexa-Vec — 1 x 10E^9 pfu (DL 2) via intravenous (IV) infusion for 4 doses: Day 12, Day 2, Day 16 of Cycle 1 and Day 2 of Cycle 2.
  Other Names: Pexa-Vec, INN pexastimogene devacirepvec
  Arms: 2/Arm A2 Pexa-Vec +Durvalumab; 4/Arm B2

SUMMARY:
Background:

* Immune-based approaches in colorectal cancer have unfortunately with the notable exception of immune checkpoint inhibition in microsatellite instable (MSI-hi) disease been largely unsuccessful. The reasons for this are unclear but no doubt relate to the fact that in advanced disease colorectal cancer appears to be less immunogenic, as evidenced by the lack of infiltrating lymphocytes with advancing T stage
* Pexa-Vec (JX-594) is a thymidine kinase gene-inactivated oncolytic vaccinia virus engineered for the expression of transgenes encoding human granulocyte- macrophage colony-stimulating factor (GM-CSF) and beta-galactosidase. Apart from the direct oncolytic activity, oncolytic viruses such as Pexa-Vec have been shown to mediate tumor cell death via the induction of innate and adaptive immune responses
* Tremelimumab is a fully human monoclonal antibody that binds to cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) expressed on the surface of activated T lymphocytes and causes inhibition of B7-CTLA-4-mediated downregulation of T-cell activation. Durvalumab is a human monoclonal antibody directed against programmed death-ligand 1 (PD-L1).
* The aim of the study is to evaluate whether the anti-tumor immunity induced by Pexa-Vec oncolytic viral therapy can be enhanced by immune checkpoint inhibition.

Objective:

-To determine the safety, tolerability and feasibility of Pexa-Vec oncolytic virus in combination with immune checkpoint inhibition in patients with refractory metastatic colorectal cancer.

Eligibility:

* Histologically confirmed metastatic colorectal cancer.
* Patients must have progressed on, been intolerant of or refused prior oxaliplatin- and irinotecan-containing, fluorouracil-based, chemotherapeutic regimen and have disease that is not amenable to potentially curative resection. Patients who have a known Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type tumor must have progressed, been intolerant of or refused cetuximab or panitumumab based chemotherapy.
* Patients tumors must be documented to be microsatellite-stable (MSS) either by genetic analysis or immunohistochemistry OR microsatellite-high with documented disease progression following anti-programmed cell death protein 1 (PD1)/Programmed death-ligand 1 (PDL1) therapy.
* Patients must have at least one focus of metastatic disease that is amenable to pre- and on-treatment biopsy.
* Willingness to undergo mandatory tumor biopsy.

Design:

-The proposed study is Phase I/II study of Pexa-Vec oncolytic virus at two dose levels in combination with immune checkpoint inhibition in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Background:

* Immune-based approaches in colorectal cancer have unfortunately with the notable exception of immune checkpoint inhibition in microsatellite instable (MSI-hi) disease been largely unsuccessful. The reasons for this are unclear but no doubt relate to the fact that in advanced disease colorectal cancer appears to be less immunogenic, as evidenced by the lack of infiltrating lymphocytes with advancing T stage
* Pexa-Vec (JX-594) is a thymidine kinase gene-inactivated oncolytic vaccinia virus engineered for the expression of transgenes encoding human granulocyte- macrophage colony-stimulating factor (GM-CSF) and beta-galactosidase. Apart from the direct oncolytic activity, oncolytic viruses such as Pexa-Vec have been shown to mediate tumor cell death via the induction of innate and adaptive immune responses
* Tremelimumab is a fully human monoclonal antibody that binds to cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) expressed on the surface of activated T lymphocytes and causes inhibition of B7-CTLA-4-mediated downregulation of T-cell activation. Durvalumab is a human monoclonal antibody directed against programmed death-ligand 1 (PD-L1).
* The aim of the study is to evaluate whether the anti-tumor immunity induced by Pexa-Vec oncolytic viral therapy can be enhanced by immune checkpoint inhibition.

Objective:

-To determine the safety, tolerability and feasibility of Pexa-Vec oncolytic virus in combination with immune checkpoint inhibition in patients with refractory metastatic colorectal cancer.

Eligibility:

* Histologically confirmed metastatic colorectal cancer.
* Patients must have progressed on, been intolerant of or refused prior oxaliplatin- and irinotecan-containing, fluorouracil-based, chemotherapeutic regimen and have disease that is not amenable to potentially curative resection. Patients who have a known Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type tumor must have progressed, been intolerant of or refused cetuximab or panitumumab based chemotherapy.
* Patient's tumors must be documented to be microsatellite-stable (MSS) either by genetic analysis or immunohistochemistry OR microsatellite-high with documented disease progression following anti-programmed cell death protein 1 (PD1)/Programmed death-ligand 1 (PDL1) therapy.
* Patients must have at least one focus of metastatic disease that is amenable to pre- and on-treatment biopsy.
* Willingness to undergo mandatory tumor biopsy.

Design:

* The proposed study is Phase I/II study of Pexa-Vec oncolytic virus at two dose levels in combination with immune checkpoint inhibition in patients with metastatic colorectal cancer.
* Patients will receive Pexa-Vec, administered intravenous (IV) every 2 weeks for 4 doses, in 4 separate arms A1, A2, B1, and B2. The first administration will be on Day (minus) 12, followed by administration on Days 2, 16 and 30 (i.e. 4 doses in total).

  * Arms A1 and A2: In addition to the oncolytic virus patients will also receive durvalumab at a flat dose of 1500 mg beginning on Day 1 followed by q28days until off-treatment criteria are met.
  * Arms B1 and B2: In addition to the oncolytic virus patients will also receive tremelimumab 300 mg and durvalumab 1500 mg on Day 1 followed by q28days subsequent continuation of the durvalumab alone until off-treatment criteria are met.
* All patients will undergo a baseline tumor biopsy and a post treatment biopsy.
* Accrual ceiling will be set at 35 to allow for patients replaceable for reasons other than toxicity.
* Patients will be restaged every 8 weeks +/- 3 days

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of Colorectal Carcinoma (CRC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study.
* Patients must have progressed on, been intolerant of or refused prior oxaliplatin- and irinotecan-containing, fluorouracil-based, chemotherapeutic regimen and have disease that is not amenable to potentially curative resection. Patients who have a known Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type tumor must have progressed, been intolerant of or refused cetuximab or panitumumab-based chemotherapy.
* Patient's tumors must be documented to be microsatellite-stable (MSS) either by genetic analysis or immunohistochemistry OR microsatellite-high with documented disease progression following anti-Programmed cell death protein 1 (PD1)/Programmed death-ligand 1 (PDL1) therapy.
* Patients must have at least one focus of metastatic disease that is amenable to pre- and on-treatment biopsy and be willing to undergo this. Ideally the biopsied lesion should not be one of the target measurable lesions, although this can be up to the discretion of the investigators.
* All patients enrolled will be required to have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of Pexa-Vec in combination with tremelimumab and/or durvalumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have acceptable organ and marrow function as defined below:

  * Leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * Platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 1.5X institution upper limit of normal
  * Hemoglobin (Hb) > 9g/dl
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) less than or equal to 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be less than or equal to 5x upper limit of normal (ULN)
  * Creatinine <1.5X institution upper limit of normal, OR
  * creatinine clearance greater than or equal to 45 mL/min/1.73 m(2), as calculated below, for patients with creatinine levels above institutional normal
* Patient must be able to understand and willing to sign a written informed consent document
* The effects of Pexa-Vec, durvalumab and tremelimumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and up to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women greater than or equal to 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Body weight >35kg

EXCLUSION CRITERIA:

* Patients who have had anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigation agents), large field radiotherapy, or major surgery must wait 4 weeks after completing treatment prior to entering the study.
* No prior exposure to immune-mediated therapy including, but not limited to, other anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, including therapeutic anticancer vaccines. The exception to this is those whose tumors are MSI-hi and are refractory to anti-PD1 monotherapy.
* Involvement in the planning and/or conduct of the study
* Previous IP assignment in the present study
* Patients who are receiving any other investigational agents.
* Inability to suspend treatment with anti-hypertensive medication (including but not limited to: diuretics, beta-blockers, angiotensin converting enzyme [ACE] inhibitors, aldosterone antagonists, etc.) for 48 hours pre and post each Pexa-Vec administration.
* Patients with severe hypertension who in the opinion of the investigator cannot withhold antihypertensive medication for 48 hours pre and post Pexa-Vec administration.
* Any unresolved toxicity NCI Common Terminology Criteria for Adverse Events (CTCAE) Grade greater than or equal to 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with Grade greater than or equal to 2 neuropathy will be evaluated on a case-by-case basis
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, hypertension (systolic blood pressure (BP) > 160, diastolic BP > 100), ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes or psychiatric illness/social situations that would limit compliance with study requirements. For patients with a history of cardiovascular disease, cardiology consultation. Echocardiogram, troponin and creatinine clearance must be obtained prior to enrollment. NOTE: Patients with active cardiac disease (e.g. myocarditis and myocardial infarction) within 12 months of study entry are excluded from study participation.
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and the investigational agent. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that Durvalumab or Tremelimumab may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events.
* Known significant immunodeficiency due to underlying illness (e.g. HIV/Acquired immunodeficiency syndrome (AIDS) and/or immune-suppressive medication including high-dose corticosteroids (defined as greater than or equal to 20 mg/day prednisone or equivalent which is ongoing at the time of enrollment and/or was taken for more than 4 weeks within the preceding 2 months of enrollment)
* History of chronic autoimmune disease (e.g. systemic lupus erythematosus or Wegener's granulomatosis, Addison's disease, multiple sclerosis, Graves' disease, Hashimoto's thyroiditis, hypophysitis, etc.) with symptomatic disease within the 3 years before enrollment. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion. In addition, a past history of certain autoimmunity e.g. rheumatoid arthritis or thyroiditis may be allowed per principal investigator (PI) discretion provided it has been quiescent for a minimum of three years. The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included
  5. Patients with celiac disease controlled by diet alone
  6. Active or history of inflammatory bowel disease (colitis, Crohn's), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea.
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing (if clinically indicated), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for hepatitis C virus (HCV) ribonucleic acid (RNA).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. computed tomography (CT) scan premedication)
  * Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note:

Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

* Female patients who are breastfeeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Pexa-Vec, breastfeeding should be discontinued if the mother is treated with Pexa-Vec. These potential risks may also apply to other agents used in this study.
* Known allergy or hypersensitivity to IP
* Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* History of sarcoidosis syndrome
* Mean QT interval corrected for heart rate (QTc) greater than or equal to 470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Patients with a history of Interstitial lung disease or pneumonitis
* Subjects with uncontrolled seizures
* History of leptomeningeal carcinomatosis
* History of hypersensitivity reaction to human or mouse antibody products.
* Patients with unhealed surgical wounds for more than 30 days
* Ongoing severe inflammatory skin condition (as determined by the Investigator) requiring medical treatment
* History of severe eczema (as determined by the Investigator) requiring medical treatment
* Patients with tumor(s) invading a major vascular structure (e.g. carotid artery) or other key anatomical structure (e.g. pulmonary airway) in the event of post treatment tumor swelling and/or necrosis (hepatic and portal vein involvement allowed)
* Patients with liver tumors in a location that would potentially result in significant clinical adverse effects in the opinion of investigator if post-treatment tumor swelling were to occur, including at the site of the common bile duct
* Clinically significant and/or rapidly accumulating ascites, pericardial and/or pleural effusions. Mild ascites that does not preclude safe tumor biopsy as protocol specified is allowed at the discretion of the treating physician.
* Medical conditions, per the investigator's judgment, that predispose the patient to untoward medical risk in the event of volume loading (e.g. intravenous [IV] fluid bolus infusion), tachycardia, or hypotension during or following treatment with Pexa-Vec
* Any prior or planned organ transplant (e.g. liver transplant)
* Patients who experienced a severe systemic reaction or side-effect as a result of a previous vaccination with vaccinia
* Pulse oximetry oxygen (O2) saturation <90% at rest on room air

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Rajani KR, Vile RG. Harnessing the Power of Onco-Immunotherapy with Checkpoint Inhibitors. Viruses. 2015 Nov 13;7(11):5889-901. doi: 10.3390/v7112914. PMID 26580645
- [Background] Kohlhapp FJ, Kaufman HL. Molecular Pathways: Mechanism of Action for Talimogene Laherparepvec, a New Oncolytic Virus Immunotherapy. Clin Cancer Res. 2016 Mar 1;22(5):1048-54. doi: 10.1158/1078-0432.CCR-15-2667. Epub 2015 Dec 30. PMID 26719429
- [Background] Heo J, Reid T, Ruo L, Breitbach CJ, Rose S, Bloomston M, Cho M, Lim HY, Chung HC, Kim CW, Burke J, Lencioni R, Hickman T, Moon A, Lee YS, Kim MK, Daneshmand M, Dubois K, Longpre L, Ngo M, Rooney C, Bell JC, Rhee BG, Patt R, Hwang TH, Kirn DH. Randomized dose-finding clinical trial of oncolytic immunotherapeutic vaccinia JX-594 in liver cancer. Nat Med. 2013 Mar;19(3):329-36. doi: 10.1038/nm.3089. Epub 2013 Feb 10. PMID 23396206
- [Derived] Monge C, Xie C, Myojin Y, Coffman K, Hrones DM, Wang S, Hernandez JM, Wood BJ, Levy EB, Juburi I, Hewitt SM, Kleiner DE, Steinberg SM, Figg WD, Redd B, Homan P, Cam M, Ruf B, Duffy AG, Greten TF. Phase I/II study of PexaVec in combination with immune checkpoint inhibition in refractory metastatic colorectal cancer. J Immunother Cancer. 2023 Feb;11(2):e005640. doi: 10.1136/jitc-2022-005640. PMID 36754451
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0092.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg: Cohort A/Dose Level 1 Durvalumab 1500mg every(q) 28 day(d); Pexa-Vec 3 x 10^8/plaque-forming unit(pfu)
- 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg: Cohort A/Dose Level 2 Durvalumab 1500mg every(q) 28 day(d); Pexa-Vec 1 x 10^9/plaque-forming unit(pfu)
- 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg: Cohort B/Dose Level 1 Tremelimumab 300mg 1x; Durvalumab 1500mg every(q) 28 day(d); Pexa-Vec 3 x 10^8/plaque-forming unit(pfu)
- 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg: Cohort B/Dose Level 2 Tremelimumab 300mg; Durvalumab 1500mg every(q) 28 day(d); Pexa-Vec 1 x 10^9/plaque-forming unit(pfu)
Period: Overall Study
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Started | 4 | 12 | 4 | 14
Completed | 3 | 11 | 0 | 14
Not Completed | 1 | 1 | 4 | 0
Not completed — Participant Noncompliance | 0 | 1 | 0 | 0
Not completed — Unable to complete the dose limiting toxicity period | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Taken off active treatment | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | Total
Number analyzed (Participants) | 4 | 12 | 4 | 14 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 3 | 12 | 28
  >=65 years | 0 | 3 | 1 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.46 (5.38) | 56.17 (10.29) | 55.89 (12.87) | 54.93 (12.66) | 54.39 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 1 | 9 | 20
  Male | 2 | 4 | 3 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 11 | 4 | 12 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 4 | 1 | 3 | 8
  White | 2 | 8 | 3 | 9 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 12 | 4 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 1-5 Adverse Events
Description: Number of participants with Grade 1-5 Adverse events. Grade 1 is mild, Grade 2 is moderate, Grade 3 severe or medically significant, Grade 4 is life-threatening consequences, and Grade 5 is death related to adverse event.
Time Frame: 30 days after last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Number analyzed (Participants) | 4 | 12 | 4 | 14
Participants
  Grade 1 | 4 | 12 | 4 | 13
  Grade 2 | 4 | 12 | 4 | 14
  Grade 3 | 4 | 9 | 3 | 10
  Grade 4 | 1 | 2 | 2 | 3
  Grade 5 | 1 | 1 | 1 | 1

2. Secondary Outcome: Percentage of Participants With 5 Month Progression-free Survival
Description: Median amount of time subject survives without disease progression after treatment at 5 months. Disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: 5 months
Measure: Number; unit: percentage of participants
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Number analyzed (Participants) | 4 | 12 | 4 | 14
percentage of participants | 0 | 8.3 | 0 | 7.1

3. Secondary Outcome: Overall Progression-free Survival
Description: Median amount of time subject survives without disease progression after treatment. Disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: At progression, approximately 9 months
Measure: Median (Full Range); unit: Months
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Number analyzed (Participants) | 4 | 12 | 4 | 14
Months | 3 [0.8 to 3.2] | 2.3 [1.3 to 9.6] | 2.25 [1.1 to 2.8] | 1.65 [0.2 to 5.5]

4. Secondary Outcome: Overall Survival
Description: Median amount of time subject survives after therapy.
Time Frame: Death, an average of 9 months
Measure: Median (Full Range); unit: Months
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Number analyzed (Participants) | 4 | 12 | 4 | 14
Months | 6.2 [1.1 to 17.3] | 8.6 [3.7 to 26.3] | 6.0 [1.1 to 12.4] | 5.2 [2.1 to 18.8]

5. Secondary Outcome: Number of Participants With Response
Description: Changes in tumor size and occurrence of metastases was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). And Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Every 2 months until disease progression or intolerable toxicity, approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Number analyzed (Participants) | 4 | 12 | 4 | 14
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 0 | 0
  Stable Disease | 0 | 0 | 1 | 1
  Progressive Disease | 3 | 10 | 2 | 9
  Unevaluable | 1 | 1 | 1 | 4

6. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.3)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.3). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 20 months and 3 days for 1/Arm A1, 30 months and 27 days for 2/Arm A2, 14 months for 3/Arm B1, and 13 months and 21 days for 4/Arm B2.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
Number analyzed (Participants) | 4 | 12 | 4 | 14
Participants | 4 | 12 | 4 | 14

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 20 months and 3 days for 1/Arm A1, 30 months and 27 days for 2/Arm A2, 14 months for 3/Arm B1, and 13 months and 21 days for 4/Arm B2.
Arm/Group | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg
All-Cause Mortality (participants affected / at risk) | 4/4 | 11/12 | 4/4 | 10/14
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/12 | 3/4 | 6/14
Other Adverse Events (participants affected / at risk) | 4/4 | 12/12 | 4/4 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg (N=4) | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg (N=12) | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg (N=4) | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg (N=14)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, immune mediated colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm A1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg (N=4) | 2/Arm A2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) +Durvalumab 1500 mg (N=12) | 3/Arm B1 Pexa-Vec 3 x 10E^8 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg (N=4) | 4/Arm B2 Pexa-Vec 1 x 10E^9 Plaque-forming Unit (Pfu) + Durvalumab 1500 mg +Tremelimumab 300 mg (N=14)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4) | 2 (5) | 4 (5)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 7 (12) | 3 (7) | 3 (6)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (5) | 5 (8) | 1 (2) | 5 (8)
Alkaline phosphatase increased (Investigations) | 1 (2) | 6 (14) | 3 (4) | 7 (11)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (9) | 12 (42) | 4 (8) | 10 (36)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 3 (4) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (6) | 6 (9) | 3 (5) | 7 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 1 (1) | 5 (8)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2) | 2 (5) | 1 (3) | 4 (13)
Chills (General disorders) | 3 (6) | 9 (23) | 4 (8) | 13 (34)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 7 (7) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 4 (11) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 3 (6)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (6)
Eye disorders - Other, Black dots in vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 8 (11) | 4 (4) | 6 (7)
Fever (General disorders) | 4 (14) | 12 (62) | 4 (14) | 13 (48)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (2) | 3 (4) | 1 (1) | 6 (10)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Abdominal Cramping (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Cramp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (7) | 0 (0) | 8 (11)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 1 (1) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 6 (13) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (4) | 2 (5) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 4 (10) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 9 (20) | 3 (8) | 8 (20)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (2) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (2) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 7 (13) | 2 (3) | 6 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 3 (7) | 3 (4)
Hypotension (Vascular disorders) | 2 (3) | 10 (23) | 1 (2) | 8 (15)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, E/coli in stool (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 3 (5)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (9) | 9 (30) | 4 (10) | 9 (26)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (6) | 5 (9) | 4 (4) | 11 (23)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1) | 4 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 2 (8) | 1 (2) | 7 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 4 (4) | 3 (3) | 3 (3)
Psychiatric disorders - Other, Somnolent (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Mucous Plug (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 2 (4) | 2 (2) | 2 (5)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 6 (14) | 2 (4) | 11 (36)
Skin and subcutaneous tissue disorders - Other, Blister - toe (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Cold sore- left lip (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Swelling - leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Vesicle (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0
Skin and subcutaneous tissue disorders - Other, bump on clavicle (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 4 (5) | 3 (4) | 10 (16)
Weight loss (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (3) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03206073/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03206073/ICF_001.pdf